CLINICAL TRIAL: NCT00839007
Title: A Multi-Center, Single-Blind, Placebo-Controlled Phase 2 Study Assessing the Safety and Efficacy of Intravenous CD-NP in the Treatment of Patients With Acute Decompensated Heart Failure
Brief Title: Study to Assess the Safety and Efficacy of CD-NP in the Treatment of Patients With Acute Decompensated Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nile Therapeutics (Industry)
Responsible Party: Hsiao Lieu, MD, Vice President, Clinical Research, Nile Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIL-CDNP-CT005
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2010-09

CONDITIONS: Acute Decompensated Heart Failure
Keywords: ADHF; AHF; HF

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- A (Experimental): Dose 1 of CD-NP
  Interventions: Drug: CD-NP
- B (Experimental): Dose 2 of CD-NP
  Interventions: Drug: CD-NP
- C (Experimental): Dose 3 of CD-NP
  Interventions: Drug: CD-NP
- D (Experimental): Dose 4 of CD-NP
  Interventions: Drug: CD-NP
- E (Experimental): Dose 5 of CD-NP
  Interventions: Drug: CD-NP
- F (Experimental): Dose 6 of CD-NP
  Interventions: Drug: CD-NP
- G (Placebo Comparator): Placebo
  Interventions: Drug: CD-NP

INTERVENTIONS:
Drug: CD-NP — Infusion of CD-NP at one of up to 6 doses or placebo

SUMMARY:
The primary objective of the study is to assess the safety and tolerability of IV administration of CD-NP and the dose relationship of CD-NP on improvement of clinical symptoms and renal function in ADHF patients.

ELIGIBILITY:
Key Inclusion Criteria:

1. Hospitalized for acute decompensated heart failure.
2. Systolic blood pressure ≥ 115 mmHg and ≤ 200 mmHg, and diastolic blood pressure ≥ 60 mmHg and ≤ 110 mmHg at screening
3. Renally compromised.
4. Female patients must be post-menopausal or surgically sterile.

Key Exclusion Criteria:

1. Acute or suspected acute myocardial infarction (AMI) or troponin levels > 3X the upper limit of normal at the institution's local laboratory
2. Cardiogenic shock
3. Evidence of uncorrected volume or sodium depletion other clinical condition that would predispose the patient to adverse events
4. Clinically significant aortic or mitral valve stenosis
5. Temperature >38°C (oral or equivalent), sepsis or active infection requiring IV anti-microbial treatment
6. ADHF due to significant arrhythmias
7. Severe renal failure defined as creatinine clearance < 30 mL/min
8. Current or planned ultrafiltration, hemofiltration, or dialysis
9. Significant pulmonary disease
10. Major neurologic event, including cerebrovascular events in the prior 60 days.
11. Acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (not including restrictive mitral filling patterns)
12. Known hypersensitivity or allergy to natriuretic peptide or its components, nesiritide, other natriuretic peptides or related compounds

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The occurence of hypotensive events, clinical symptoms, and renal function change with CD-NP infusion. | Up to 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao Lieu, MD, Study Director — Nile Therapeutics
Locations (20):
- United States (10):
  - Los Angeles, California
  - Torrance, California
  - Jacksonville, Florida
  - Miami Beach, Florida
  - Chicago, Illinois
  - Iowa City, Iowa
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - The Bronx, New York
  - Houston, Texas
- Germany (4):
  - Berlin
  - Dortmund
  - Neuss
  - Würzberg
- Israel (6):
  - Ashkelon
  - Haifa
  - Nazareth
  - Petah Tikva
  - Safed
  - Tel Aviv